CLINICAL TRIAL: NCT02283853
Title: Open-Label, Randomized, Multicenter, Multiple-Dose,Active-Controlled, Parallel-Group, Efficacy and Safety Study of BG00012 in Children From 10 to Less Than 18 Years of Age With Relapsing-Remitting Multiple Sclerosis, With Optional Open-Label Extension
Brief Title: Phase 3 Efficacy and Safety Study of BG00012 in Pediatric Subjects With Relapsing-remitting Multiple Sclerosis (RRMS)
Acronym: CONNECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 109MS306; 2013-002318-11 (EudraCT Number)
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Pediatrics
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Dimethyl Fumarate; Interferon beta-1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- BG00012 (Experimental): Participants will receive the recommended dose of 240 mg orally, twice a day
  Interventions: Drug: dimethyl fumarate
- IFN β-1a (Avonex) (Active Comparator): Participants will receive the recommended dose of 30 μg (weekly)
  Interventions: Drug: Interferon β-1a

INTERVENTIONS:
Drug: dimethyl fumarate — administered orally
  Other Names: BG00012; Tecfidera
  Arms: BG00012
Drug: Interferon β-1a — administered by intramuscular injection
  Other Names: Avonex
  Arms: IFN β-1a (Avonex)

SUMMARY:
The main objectives of Part 1 are as follows: To evaluate the safety, tolerability, and efficacy of BG00012 in pediatric subjects with RRMS, as compared with a disease-modifying treatment and to assess health outcomes and evolution of disability. The primary objective of Part 2 is to evaluate the long-term safety of BG00012 in subjects who completed Week 96 in Part 1 of Study 109MS306. The secondary objective of Part 2 is to describe the long-term MS outcomes of BG00012 in subjects who completed Week 96 in Part 1 of Study 109MS306.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have a body weight of ≥30 kg.
* Must have a diagnosis of RRMS (consensus definition for pediatric RRMS [Krupp 2007]).
* Must be ambulatory with a baseline EDSS score between 0 and 5.5, inclusive.
* Must have experienced at least 1 of the following 3 conditions: a) at least 1 relapse within the last 12 months prior to Day 1 with a prior brain MRI demonstrating lesions consistent with MS; b) at least 2 relapses within the last 24 months prior to Day 1, with a prior brain MRI demonstrating lesions consistent with MS; c) evidence of Gd-enhancing lesions of the brain on an MRI performed within the 6 weeks prior to Day 1.
* Must be neurologically stable, with no evidence of relapse within 50 days prior to Day 1 and no evidence of corticosteroid treatment within 30 days prior to Day 1.
* Subjects of childbearing potential who are sexually active must be willing to practice effective contraception during the study and be willing and able to continue contraception for at least 30 days after their final dose of study treatment.

Key Exclusion Criteria:

* Primary progressive, secondary progressive, or progressive relapsing MS (as defined by [Lublin and Reingold 1996]). These conditions require the presence of continuous clinical disease worsening over a period of at least 3 months. Subjects with these conditions may also have superimposed relapses but are distinguished from relapsing-remitting subjects by the lack of clinically stable periods or clinical improvement.
* Disorders mimicking MS, such as other demyelinating disorders (e.g., acute disseminated encephalomyelitis), systemic autoimmune disorders (e.g., Sjögren disease, lupus erythematosus), metabolic disorders (e.g., dystrophies), and infectious disorders.
* History of premalignant or malignant disease. Subjects with basal cell carcinoma that has been completely excised prior to screening will remain eligible.
* History of severe allergic or anaphylactic reactions, or known drug hypersensitivity to DMF, fumaric acid esters, or interferon beta-1a (IFN Beta-1a).
* History of abnormal laboratory results indicative of any significant endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, renal, and/or any other major disease that would preclude participation in a clinical study.
* History of clinically significant cardiovascular, pulmonary, GI, dermatologic, growth, developmental, psychiatric (including depression), neurologic (other than MS), and/or other major disease that would preclude participation in a clinical study.

  -.History of human immunodeficiency virus.
* An MS relapse that has occurred within 50 days prior to Day 1 AND/OR the subject has not stabilized from a previous relapse prior to Day 1.
* Other unspecified reasons that, in the opinion of the Investigator or Biogen Idec, make the subject unsuitable for enrollment.
* For the PD/PK subset of subjects: subjects unable to swallow the BG00012 capsule whole.

Key Treatment history

* Any previous treatment with Fumaderm (fumaric acid esters) or BG00012.
* Prior treatment with any of the following: total lymphoid irradiation, cladribine, T-cell or T-cell receptor vaccination, any therapeutic monoclonal antibody, with the exception of rituximab or natalizumab.
* Prior treatment with any of the following medications within the 12 months prior to Day 1: mitoxantrone, cyclophosphamide, rituximab.
* Prior treatment with any of the following medications or procedures within 6 months prior to Day 1: fingolimod; teriflunomide; natalizumab; cyclosporine; azathioprine; methotrexate; mycophenolate mofetil; laquinimod; intravenous (IV) immunoglobulin; plasmapheresis or cytapheresis
* Treatment with any of the following medications within 30 days prior to Day 1: steroids (IV or oral corticosteroid treatment, including agents that may not act through the corticosteroid pathway [e.g.low dose naltrexone]), 4-aminopyridine or related products (except subjects on a stable dose of controlled-release fampridine for 3 months)

NOTE: Other protocol-defined inclusion/exclusion criteria may apply

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 156 (Actual)
Dates: Start 2014-08-28 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants Free of New/Newly Enlarging T2 Hyperintense Lesions on Brain MRI Scans | At week 96
  Part 1
Number of Participants That Experience Adverse Events (AEs) or Serious Adverse Events (SAEs) | Up to 7 years
  Part 2 will be an optional open-label extension phase in subjects who complete Part 1 and who meet the Part 2 entry criteria.
Number of Participants Who Discontinue Study Treatment due to an AE | Up to 7 years
  Part 2

SECONDARY OUTCOMES:
The Number of New/Newly Enlarging T2 Hyperintense Lesions on Brain MRI Scans | At Week 24 and Week 96
  Part 1
Proportion of Participants Free of New/Newly Enlarging T2 Hyperintense Lesions on Brain MRI Scans | At Week 24 and Week 48
  Part 1
Proportion of Participants Free of New MRI Activity as measured by Brain MRI Scans | At Weeks 24, 48 and 96
  Part 1. New MRI Activitiy includes: Gd-enhancing MRI lesions on brain MRI scans; New T2 MRI lesions on brain MRI scans and newly enlarging MRI lesions on brain MRI scans
Time to First Relapse | Up to Week 96
  Part 1
Proportion of Participants Who Do Not Experience Relapse | Up to Week 96
  Part 1
Annualized Relapse Rate | At Weeks 48 and 96
  Part 1
Number of Participants That Experience Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Week 96
  Part 1. Including prospective and follow-up of flushing, nausea, abdominal pain and diarrhea
Fatigue as measured by the Pediatric Quality of Life Inventory (PedsQL) Multidimensional Fatigue Scale Scores | Up to Week 96
  Part 1. Multidimensional Fatigue Scale scores - designed as a generic symptom-speciﬁc instrument to measure fatigue in patients with acute and chronic health conditions as well as healthy school and community populations.
Quality of Life as measured by the PedsQL | Up to Week 96
  Part 1
Change from Baseline to Week 96 in the Expanded Disability Status Scale (EDSS) Score | Up to Week 96
  Part 1. The EDSS measures the disability status of people with multiple sclerosis on a scale that ranges from 0 to 10. The first levels 1.0 to 4.5 refer to people with a high degree of ambulatory ability and the subsequent levels 5.0 to 9.5 refer to the loss of ambulatory ability. The range of main categories include (0) = normal neurologic exam; to (5) = ambulatory without aid or rest for 200 meters; disability severe enough to impair full daily activities; to (10) = death due to MS.
Vital Signs, Electrocardiograms (ECGs) and Changes in Clinical Laboratory Data, including Monitoring of Liver Function, Renal Function, Hematologic, and Coagulation Parameters | Up to Week 96
  Part 1
Annualized Relapse Rate | Up to 7 years
  Part 2
Change from Baseline in EDSS Score | Up to 7 years
  Part 2. The EDSS measures the disability status of people with multiple sclerosis on a scale that ranges from 0 to 10. The first levels 1.0 to 4.5 refer to people with a high degree of ambulatory ability and the subsequent levels 5.0 to 9.5 refer to the loss of ambulatory ability. The range of main categories include (0) = normal neurologic exam; to (5) = ambulatory without aid or rest for 200 meters; disability severe enough to impair full daily activities; to (10) = death due to MS.
Change from Baseline in Symbol Digit Modalities Test (SDMT) Score | Up to 7 years
  Part 2. SDMT is used to assess processing speed. Participants are given 90 seconds in which to pair specific numbers with given geometric figures using a key. The score is number of correctly coded items from 0 (worst) to 110 (best). Higher scores indicate better performance.
Change from Baseline in Brief Visuospatial Memory Test - Revised (BVMT-R) Score | Up to 7 years
  Part 2. BVMT-R is used to assess learning/memory. The stimulus page is presented for 10 seconds, and the participant is then asked to reproduce the designs as accurately as possible and in the same location on the page. Three learning trials are administered, followed by a delay trial approximately 20 to 40 minutes later. Immediately following the delay trial a recognition trial is administered to see whether the participant recognizes the figures that were on the display.
Change from Baseline in School Progression Query | Up to 7 years
  Part 2. If permitted by the local regulatory authority, participants or caregivers will be posed the following question: "During the past year, did [you/the subject] progress from one [class/grade-level] to the next in school?"
Number of Participants with Incidences of Clinically Relevant Vital Signs Abnormalities | Up to 7 years
  Part 2
Number of Participants with Incidences of Clinically Relevant ECG Abnormalities | Up to 7 years
  Part 2
Number of Participants with Incidences of Clinically Relevant Laboratory Assessment Abnormalities | Up to 7 years
  Part 2
Change from Baseline in Height | Up to 7 years
  Part 2
Change from Baseline in Weight | Up to 7 years
  Part 2
Change from Baseline in Bone Age | Up to 7 years
  Part 2
Tanner Stage | Up to 7 years
  Part 2. Information regarding Tanner staging will be collected at baseline for all male participants and for female participants who are premenarche and will be stopped once the participant's bone age reaches ≥16 years or once the participant is postmenarche.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (62):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - The Rector and Visitors of the University of Virginia, Charlottesville, Virginia
- Belgium (2):
  - Universitair Kinderziekenhuis Koningin Fabiola, Brussels
  - Universitair Ziekenhuis Ghent, Ghent
- MHATNP 'Sv.Naum', EAD, Sofia, Bulgaria
- University of Calgary - Alberta Children's Hospital, Calgary, Alberta, Canada
- Czechia (4):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Nemocnice Jihlava p.o., Jihlava
  - Fakultni nemocnice Ostrava, Ostrava
- Denmark (3):
  - Århus Universitetshospital, Aarhus N
  - Rigshospitalet, Copenhagen
  - Odense Universitetshospital, Odense
- France (11):
  - CHU Strasbourg - Hôpital Hautepierre, Strasbourg, Bas Rhin
  - Hôpital de la Timone, Marseille, Bouches-du-Rhône
  - CHU Dijon -BOCAGE CENTRAL, Dijon, Côte-d'Or
  - Hopital Gui de Chauliac, Montpellier, Herault
  - CHU Rennes - Hopital Pontchaillou, Rennes, Ille Et Vilaine
  - Hôpital de Brabois Enfants, Vandœuvre-lès-Nancy, Meurthe Et Moselle
  - Hopital Roger Salengro - CHU Lille, Lille, Nord
  - CHU Clermont Ferrand - Hôpital d'Estaing, Clermont-Ferrand, Puy De Dome
  - Hopital Neurologique Pierre Wertheimer, Bron, Rhone
  - CHU Amiens - Hopital Sud, Amiens, Somme
  - Hôpital Bicêtre, Le Kremlin-Bicêtre, Val De Marne
- Germany (3):
  - Universitaetsklinikum Augsburg, Augsburg, Bavaria
  - Klinikum der Universitaet Muenchen, Munich, Bavaria
  - Katholisches Klinikum Bochum gGmbH, Bochum, North Rhine-Westphalia
- Hungary (2):
  - Semmelweis Egyetem, Budapest
  - Heim Pal Orszagos Gyermekgyogyaszati Intezet, Budapest
- Israel (3):
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Schneider Children's Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
- Italy (9):
  - Azienda Socio Sanitaria Territoriale della Valle Olona (presidio di Gallarate), Gallarate, Varese
  - Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliera Universitaria 'Federico II', Napoli
  - Azienda Ospedale-Università di Padova, Padua
  - Azienda Ospedaliero Universitaria Policlinico Paolo Giaccone, Palermo
  - Ospedale Pediatrico Bambino Gesù, Roma
  - Azienda Ospedaliera Sant'Andrea-Università di Roma La Sapienza, Roma
- Ibn Sina Hospital, Ash Shuwaykh, Kuwait
- Poland (5):
  - SPZOZ Uniwersytecki Dzieciecy Szpital Kliniczny im. L. Zamenhofa, Bialystok
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Szpital Kliniczny im.Heliodora Swiecickiego Uniwersytetu Medycznego im.K. Marcinkowskiego w Poznaniu, Poznan
  - Instytut 'Pomnik - Centrum Zdrowia Dziecka', Warsaw
- Serbia (3):
  - Clinic of Neurology and Psychiatry for Children and Youth, Belgrade
  - Mother and Child Health Care Institute of Serbia ,,Dr Vukan Cupic'', Belgrade
  - University Clinical Center Kragujevac, Kragujevac
- Spain (4):
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba, Córdoba
  - Hospital Universitario de Torrejon, Torrejón de Ardoz, Madrid
  - Hospital Universitario Virgen Macarena, Seville
- Sweden (2):
  - Sahlgrenska Sjukhuset, Gothenburg
  - Karolinska, Stockholm
- Turkey (Türkiye) (2):
  - Hacettepe University Medical Faculty, Ankara
  - Akdeniz University Faculty of Medicine, Antalya
- United Kingdom (4):
  - Evelina London Children's Hospital, London, Greater London
  - The National Hospital for Neurology & Neurosurgery, London, Greater London
  - Great Ormond Street Hospital for Children, London, Greater London
  - Birmingham Children's Hospital, Birmingham, West Midlands

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/.
URL: https://vivli.org

REFERENCES:
- [Derived] Vermersch P, Scaramozza M, Levin S, Alroughani R, Deiva K, Pozzilli C, Lyons J, Mokliatchouk O, Pultz J, N'Dure F, Liu S, Badwan R, Branco F, Hood-Humphrey V, Franchimont N, Hanna J, Maghzi AH. Effect of Dimethyl Fumarate vs Interferon beta-1a in Patients With Pediatric-Onset Multiple Sclerosis: The CONNECT Randomized Clinical Trial. JAMA Netw Open. 2022 Sep 1;5(9):e2230439. doi: 10.1001/jamanetworkopen.2022.30439. PMID 36169959